CLINICAL TRIAL: NCT04750798
Title: An Observational Post-marketing Study for Evaluation of Ongoing Safety and Effectiveness of Catheter Mapping and Ablation Using Commercially Approved BWI Medical Devices for the Treatment of Patients With Cardiac Arrhythmias
Brief Title: An Observational Post-marketing Study Using Commercially Approved Biosense Webster (BWI) Medical Devices for the Treatment of Participants With Cardiac Arrhythmias
Acronym: SECURE
Status: Recruiting | Type: Observational
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BWI_2019_05
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Participants Diagnosed with Cardiac Arrhythmias: Patients diagnosed with cardiac arrhythmias who are scheduled to undergo an ablation procedure in routine clinical practice for management of their arrhythmia with a BWI therapeutic catheter/Varipulse Catheter/ Dual Energy Thermocool Smarttouch surround flow (SF) catheter will be observed.
  Interventions: Device: BWI Medical Device; Device: Varipulse Catheter; Device: Dual Energy THERMOCOOL SMARTTOUCH SF Catheter

INTERVENTIONS:
Device: BWI Medical Device — Participants will be treated with commercially approved BWI medical devices following routine clinical practice. No specific intervention will be observed for this study.
Device: Varipulse Catheter — Participants treated with Varipulse Catheter in the main study will be part of the VARIPURE sub-study. No specific intervention will be observed for this study.
Device: Dual Energy THERMOCOOL SMARTTOUCH SF Catheter — Participants treated with the Dual Energy THERMOCOOL SMARTTOUCH SF Catheter in the main study will be part of the DUACURE sub-study. No specific intervention will be observed for this study.

SUMMARY:
The purpose of this study is to prospectively collect clinical data evaluating the ongoing safety and performance during routine-use standard cardiac arrhythmia mapping and/or ablation procedures while using commercial Biosense Webster Inc. (BWI) medical devices. Data generated from the study will be used to confirm safety and performance of BWI medical devices in the marketed phase and to expand the body of evidence on the use of these devices and techniques in treatment of cardiac arrhythmias.

ELIGIBILITY:
Inclusion criteria

* Diagnosed with paroxysmal or persistent Atrial Fibrillation (AF) or supraventricular tachycardia (SVT) or ventricular tachycardia (VT) and scheduled to undergo an ablation procedure for management of their arrhythmia with a per-protocol defined BW therapeutic catheter
* Able and willing to comply with all pre, post and follow-up testing and requirements as per hospital standard of care
* Signed patient informed consent form (ICF) as applicable per local regulation

Exclusion criteria:

* Currently participating in an interventional (drug, device, biologic) clinical trial
* Life expectancy of less than 12-months
* Presenting any contraindication for the use of BWI commercially approved medical devices, as indicated in the respective user manuals

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population consists of participants diagnosed with cardiac arrhythmias who are scheduled to undergo an ablation procedure for management of their arrhythmia with a per-protocol defined Biosense Webster Inc (BWI) therapeutic catheter.
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2036-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Primary Adverse Events (PAEs) Related to Device in Scope and/or Study Procedure Within 7 Days of the Initial Study Procedure | Up to 7 Days
  PAEs in participants with Atrial Fibrillation (AF) and for SupraVentricular Tachycardia (SVT) includes device or procedure related death, atrio-esophageal fistula/ esophageal perforation , severe pulmonary vein stenosis, cardiac tamponade/perforation, thromboembolism, pericarditis, stroke/cerebrovascular accident, transient ischemic attack, phrenic nerve paralysis (permanent), myocardial infarction, major vascular access complication/bleeding, heart block; PAEs in participants with Ventricular Tachycardia (VT) includes device or procedure related death, cardiac tamponade/perforation, thromboembolism, pericarditis, stroke/cerebrovascular accident, transient ischemic attack, phrenic nerve paralysis (permanent), myocardial infarction, major vascular access complication/bleeding, heart block, aggravation or new onset heart failure, coronary artery injury, aortic dissection and valve injury.
AF: Number of Participants with Isolation of all Targeted Pulmonary Veins | Up to 7 Days
  Number of Participants with isolation (entrance block confirmation) of all targeted pulmonary veins will be reported.
SVT (Sinus Nodal Re-entrant Tachycardia, Focal AT, Multifocal AT, AVNRT, Non Re-entrant Junctional Tachycardias): Number of Participants with Non-inducibility of the Targeted Tachycardia at end of Procedure | Up to 7 Days
  Number of participants with sinus nodal re-entrant tachycardia, focal atrial tachycardia (AT) multifocal AT, atrioventricular nodal reentry tachycardia (AVNRT), non re-entrant junctional tachycardias with non-inducibility of the targeted tachycardia at end of procedure will be reported.
SVT (MRAT): Number of Participants with Complete Bidirectional Conduction Block Across the Ablation Line | Up to 7 Days
  Number of participants with Macro Re-entrant Atrial Tachycardia (MRAT) with complete bidirectional conduction block across the ablation line will be reported.
SVT (AVRT): Number of Participants with Complete Block of Accessory Pathway | Up to 7 Days
  Number of participants with atrioventricular reentry tachycardia (AVRT) with complete block of accessory pathway will be reported.
VT (Ischemic or Non-ischemic): Number of Participants with Non-inducibility of the Targeted VT at end of Procedure | Up to 7 days
  Number of participants with non-inducibility of the targeted ischemic or non-ischemic VT at end of procedure will be reported.
VT (Idiopathic): Number of Participants with Elimination of Clinically Relevant VT | Up to 7 days
  Number of participants with elimination of clinically relevant idiopathic VT will be reported. Clinically relevant: any spontaneous VT or any induced VT.
VT (Idiopathic): Number of Participants with Elimination of Clinically Relevant Premature Ventricular Contraction (PVCs) | Up to 7 days
  Number of participants with elimination of clinically relevant idiopathic PVCs will be reported. Clinically relevant: any spontaneous PVC or any induced PVC; prior to treatment, PVCs would be deemed clinically relevant if they are present greater than (>) 20 percent (%) of daily heartbeat.

SECONDARY OUTCOMES:
Number of Participants with Device and/or Procedure-Related Serious Adverse Events (Serious Adverse Device Effects [SADEs]) | Up to 365 Days
  Number of participants with device and/or procedure-related Serious Adverse Events (SADEs) within 7 days (early-onset), >7-30 days (peri-procedural) and >30 days (late onset) following the initial study procedure will be reported.
Number of Participants with Device and/or Procedure-Related Non-Serious Adverse Events (Non-Serious Adverse Device Effects [ADEs]) | Up to 365 Days
  Number of participants with device and/or procedure-related non-serious adverse events (Non-serious ADEs) within 7 days (early-onset), >7-30 days (peri-procedural) and >30 days (Late Onset) following the initial study procedure will be reported.
AF: Number of Participants with Acute Reconnection Among all Targeted Pulmonary Veins (PVs) | Up to 7 Days
  Number of participants with Acute reconnection among all targeted PVs will be reported.
SVT (MRAT): Number of Participants with Non-inducibility of the Targeted Tachycardia at end of Procedure | Up to 7 Days
  Number of participants with MRAT with non-inducibility of the targeted tachycardia at end of procedure will be reported.
SVT (AVNRT): Number of Participants with Elimination or Modification of Slow Pathway Conduction | Up to 7 Days
  Number of participants with AVNRT with elimination or modification of slow pathway conduction will be reported.
VT (Ischemic or Non-ischemic): Number of Participants with Non-inducibility of any VT at end of Procedure | Up to 7 Days
  Number of participants with non-inducibility of any VT (Ischemic or Non-ischemic) at end of procedure will be reported.
VT (Ischemic or Non-ischemic): Number of Participants with Elimination of all Targeted Late Potentials and Local Abnormal Ventricular Activation (LAVAs) at end of Procedure | Up to 7 Days
  Number of participants with elimination of all targeted late potentials and local abnormal ventricular activation (LAVAs) at end of procedure will be reported.
AF: Number of Participants with Freedom From Documented (Symptomatic and Asymptomatic) AF, AT, Atrial Flutter (AFL) Episodes | From Day 91 to Day 365 (post-blanking)
  Number of participants with freedom from documented (symptomatic and asymptomatic) AF, AT, AFL episodes (episodes greater than or equal to [>=] 30 seconds) post-blanking will be reported.
AF: Number of Participants with Freedom From Documented Symptomatic AF, AT, AFL Episodes | From Day 91 to Day 365 (post-blanking)
  Number of participants with freedom from documented symptomatic AF, AT, AFL episodes (episodes >= 30 seconds) post-blanking will be reported.
AF: Number of Participants with Repeated Ablation | From Day 91 to Day 365 (post-blanking)
  Number of participants with repeated ablation post-blanking will be reported.
AF: Number of Participants with Repeated Ablation with Pulmonary Vein (PV) Reconnection | From Day 91 to Day 365 (post-blanking)
  Number of participants with repeated ablation with PV reconnection post blanking will be reported.
SVT: Number of Participants with Freedom From Documented Arrhythmia of the Primary SVT | From Day 1 to Day 365
  Number of participants with freedom from documented arrhythmia of the primary SVT (episodes >=30 seconds) will be reported.
SVT: Number of Participants with Freedom From Documented Arrhythmia of new SVT, not Targeted During Index Procedure | From Day 1 to Day 365
  Number of participants with freedom from documented arrhythmia of new SVT, not targeted during index procedure will be reported.
SVT: Number of Participants with Repeated Ablation | From Day 1 to Day 365
  Number of participants with repeated ablation will be reported.
VT: Number of Participants with Freedom From Documented Arrhythmia of the Clinically Relevant/Targeted VT | From Day 1 to Day 365
  Number of participants with freedom from documented arrhythmia of the clinically relevant /targeted VT (episodes >=30 seconds) will be reported.
VT: Number of Participants with Freedom From Documented Arrhythmia of new VT, not Targeted During Index Procedure | From Day 1 to Day 365
  Number of participants with freedom from documented arrhythmia of new VT, not targeted during index procedure will be reported.
VT: Number of Participants with Repeated Ablation | From Day 1 to Day 365
  Number of participants with repeated ablation will be reported.
VT: Number of Participants with All Cause and Cardiac Mortality | Up to Day 365
  Number of participants with all cause and cardiac mortality will be reported.
VT: Number of Participants with Heart Failure Hospitalization | Up to Day 365
  Number of participants with heart failure hospitalization will be reported.

OTHER OUTCOMES:
VARIPURE sub-study: Number of Participants With Coronary Spasm During Ablation | Up to Day 365
  Ablation procedures using the varipulse medical device will be performed according to the hospital standard practice. Number of participants with coronary spasm during ablation will be reported.
VARIPURE Sub-Study: Number of Participants With Vagal Response During Ablation | Up to Day 365
  Ablation procedures using the varipulse medical device will be performed according to the hospital standard practice. Number of participants with vagal response during ablation will be reported.
VARIPURE Sub-Study: Number of Participants With Acute Kidney Failure Post Ablation | Up to Day 365
  Ablation procedures using the varipulse medical device will be performed according to the hospital standard practice. Number of participants with acute kidney failure post ablation will be reported.
DUACURE Sub-Study: Number of Participants With Coronary Spasm During Ablation | Up to Day 365
  Ablation procedures using the duacure medical device will be performed according to the hospital standard practice. Number of participants with coronary spasm during ablation will be reported.
DUACURE Sub-Study: Number of Participants With Vagal Response During Ablation | Up to Day 365
  Ablation procedures using the duacure medical device will be performed according to the hospital standard practice. Number of participants with vagal response during ablation will be reported.
DUACURE Sub-Study: Number of Participants With Acute Kidney Failure Post Ablation | Up to Day 365
  Ablation procedures using the duacure medical device will be performed according to the hospital standard practice. Number of participants with acute kidney failure post ablation will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Biosense Webster, Inc. Clinical Trial, Study Director — Biosense Webster, Inc.
Locations (34):
- Austria (2):
  - Medical University of Graz, Graz
  - Ordensklinikum Linz GMBH, Linz
- Belgium (7):
  - OLV Aalst, Aalst
  - AZ Sint-Jan Brugge, Bruges
  - CHU Saint-Pierre, Brussels
  - UZ Antwerp, Edegem
  - Jessa Hospital, Hasselt
  - UZ Brussels, Jette
  - ASBL CHU HELORA Hôpital de La Louvière site Jolimont, La Louvière
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
- France (4):
  - Les Hospices Civils de Lyon, Lyon
  - Hôpital Saint Joseph de Marseille, Marseille
  - Institut Mutualiste Montsouris, Paris
  - Centre Hospitalier Universitaire de Bordeaux, Talence
- Germany (6):
  - Rhön-Klinikum Campus Bad Neustadt, Bad Neustadt an der Saale
  - Herz- und Diabeteszentrum NRW, University Hospital of the Ruhr University Bochum, Bad Oeynhausen
  - Segeberger Kliniken, Bad Segeberg
  - Alfried Krupp Hospital, Essen
  - Cardioangiologisches Centrum Bethanien (CCB), Frankfurt
  - German Heart Centre Munich, Munich
- Mater Private Heart and Vascular Centre, Dublin, Ireland
- Israel (2):
  - Shaare Zedek Medical Center, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (2):
  - Ospedale Generale Regionale "F. Miulli", Acquaviva delle Fonti
  - IRCCS Policlinico San Donato, Milan
- Netherlands (2):
  - Clinical Trial Center Maastricht, Maastricht
  - Erasmus University Medical Center, Rotterdam
- Hospital de Santa Cruz, Carnaxide, Portugal
- INSELSPITAL Universitätsspital Bern, Bern, Switzerland
- United Kingdom (4):
  - Glenfield Hospital, Leicester
  - St. Bartholomew's Hospital, London
  - St George's Hospital, London
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency